CLINICAL TRIAL: NCT07008924
Title: Partial Sleep Restriction in Chronic Low Back Pain: A Feasibility Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Neena Sharma, PT, PhD, CMPT, Associate Professor, University of Kansas Medical Center
Other Study IDs: STUDY00148602
Record Dates: First submitted 2022-07-20; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low-back Pain; Insomnia; Sleep
Keywords: Partial sleep restriction; Chronic low back pain; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Healthy control group will consist of those without any pain and sleep issues.
  Interventions: Other: No intervention is provided. We monitor natural recovery to full sleep.
- Chronic Low Back Pain (CLBP): CLBP group will consist of those with LBP. Individuals with CLBP who also experience minor sleep issues are also eligible.
  Interventions: Other: No intervention is provided. We monitor natural recovery to full sleep.

INTERVENTIONS:
Other: No intervention is provided. We monitor natural recovery to full sleep. — Return to normal sleep observation.

SUMMARY:
Our goal is to observational study is to determine feasibility of partial sleep restriction in individuals with CLBP+I and correlation findings with features of central sensitization.

* Identify feasibility of sleep restriction protocol
* Identify correlation between less sleep and central sensitization Sleep will be monitored for 2 weeks (baseline sleep monitoring period). Then participants will be asked to restrict their sleep to 80% of their normal sleep duration for 5 nights (sleep restriction period). Then sleep will be monitored again for 2 weeks (sleep recovery period).

DETAILED DESCRIPTION:
Actigraph and sleep diaries will be used to record sleep time and quality of sleep for 2 weeks baseline period. During this period several measures for pain, sleep, fatigue, cognition, and psychological status will be completed. Quantitative sensory testing will be used to establish pain threshold. Then, the participants will partial sleep restriction (20% sleep reduction/night for 5 nights). Following the completion of restricted sleep period, all outcome measures related to pain, sleep, fatigue, cognition, and psychological status will be assessed (post-sleep restriction assessment). Then participants' sleep will be monitored for 2-weeks (sleep recovery period). During the 5-night of sleep restriction, participants will be asked to complete electronic daily diary related to sleep, pain, fatigue, psychological distress and physical activity. Potential risk related to less sleep will be clearly explained to all potential individuals interested in participating.

ELIGIBILITY:
Inclusion Criteria:

• 25-65 years old individuals

Additional inclusion criteria for individuals with CLBP+I:

* With or without insomnia
* CLBP (LBP for at least 3 months with or without referred or radiating leg pain; pain intensity 1 or greater on 0 - 10 VAS scale
* likely to participate in all scheduled evaluations and study procedures by self-report
* agrees to abide by safely protocol e.g. not to drive or operate heavy machinery and perform heavy labor work, during the sleep-restriction period

Exclusion Criteria:

* spine compression, tumor, infection, history of spine surgery
* neurological conditions such as stroke, Parkinson's disease, Alzheimer's disease or other cognitive impairments.
* pregnancy
* known untreated sleep disorder (such as current sleep apnea or current restless leg syndrome) screened by the following scales to ensure insomnia symptoms are due to insomnia and not another common sleep disorders:
* Those with increased risk of sleep apnea
* Increased risk of restless leg syndrome on RLS-Diagnosis Index
* Increased risk of circadian rhythm sleep-wake disorder
* Increased risk of parasomnia
* Moderate level of depression identified by Patient Health Questionnaire (PHQ-9)
* Moderate level of anxiety identify by Generalized Anxiety Disorder (GAD-7)
* history of drug or alcohol abuse as defined by DSM-IV criteria within the last 2 years
* severe mental illness such as schizophrenia or bipolar disorder
* developmental history of learning disability or attention-deficit/hyperactivity disorder
* is currently receiving CBT-I, physical therapy or chiropractic treatment
* history of spinal surgery
* current use of blood thinning medications
* resting blood pressure greater than 160/90 mmHg40,49,50
* performs overnight shift work

Additional exclusion criteria for HC individuals:

• pain rating 0 out of 0 - 10 Numeric Rating Pain Scale in any parts of the body

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will primarily recruit patients via word of mouth, by placing study flyers throughout KU hospital and KUMC and social media e.g. broadcast, facebook, etc. We may also use KUMC's CTSA Frontiers patient registry to recruit participants with LBP. Attach is a copy of study flyer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Measures | Through study completion, up to 5 weeks
  Daily electronic sleep diaries
Sleep Measures | Through study completion, up to 5 weeks
  Insomnia Severity Index (ISI)
Sleep Measures | Through study completion, up to 5 weeks
  Pittsburgh Sleep Quality
Pain Measures | Through study completion, up to 5 weeks
  Daily pain diaries
Pain Measures | Through study completion, up to 5 weeks
  SF-McGill (MPQ),

SECONDARY OUTCOMES:
Sleep Measures | Through study completion, up to 5 weeks
  Actigraphy- wearable sensor to record sleep quality and duration.
Pain Measures | Through study completion, up to 5 weeks
  Numeric pain rating
Pain Measures | Through study completion, up to 5 weeks
  2011 FM Survey
Pain Measures | Through study completion, up to 5 weeks
  McGill pain questionnaire
Pain Measures | Through study completion, up to 5 weeks
  Pressure pain threshold (PPT), lower back and dominant thumbnail
Pain Measures | Through study completion, up to 5 weeks
  Conditioned Pain Modulation (CPM):lower back and dominant thumbnail
Pain Measures | Through study completion, up to 5 weeks
  Pinprick assessment
Psychological Measures | Through study completion, up to 5 weeks
  Beck Anxiety Index (BAI)
Psychological Measures | Through study completion, up to 5 weeks
  Beck Depression Inventory (BDI-I)
Psychological Measures | Through study completion, up to 5 weeks
  Perceived Stress Scale (PSS)
Psychological Measures | Through study completion, up to 5 weeks
  Multidimensional Fatigue Inventory (MFI)- quantify different facets of fatigue.
Psychological Measures | Through study completion, up to 5 weeks
  Catastrophizing Scale (PCS)
Daily questionnaire | Through study completion, up to 5 weeks
  For sleep restriction and recovery periods

CONTACTS AND LOCATIONS:
Overall Officials: Neena Sharma, Principal Investigator — university
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No